CLINICAL TRIAL: NCT02332525
Title: The Influence of Oral Vibrational Stimulation on Brain Activity and Cognitive Function of Elderly Individuals With Mild Cognitive Impairment
Brief Title: The Influence of Oral Vibrational Stimulation on Cognitive Function of Elderly Individuals
Acronym: OVSCF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Lee, Hyo-Jung, assistant professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1407-260-006
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Oral Vibrational Stimulation; Cognitive Function; Mild Cognitive Impairment; cognitive normal elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): 20 elders (10 mild cognitive impairment, 10 cognitive normal elders) those who received oral vibrational stimulation
  Interventions: Device: Oral Vibrational Stimulation

INTERVENTIONS:
Device: Oral Vibrational Stimulation — Oral application of vibratory stimulus
  : With the oral equipment, which is similar to the device generally used to prevent teeth grinding in dental clinics, 15-second vibratory and 15-second non-vibratory stimulus are given repeatedly for about 5 minutes using a vibrator that has a strength less than or equal to the vibratory stimulus of a smartphone (3.3V, 166Hz, maximum 180Hz). A stimulus of two times for 5 minutes, a total of at least 10 minutes is conducted for 10 days in a hospital or designated place.

SUMMARY:
The purpose of this study is to investigate the effect of oral vibratory stimulus on the brain activity and cognitive function of elderly people with non-dementia subjects (cognitive normal, mild cognitive impairment)

DETAILED DESCRIPTION:
Evaluating the effect of oral vibratory stimulus on the brain activity and cognitive function of elderly people with mild cognitive impairment

◇ Test design: Open-labeled, prospective, pre-post study

○ Oral vibratory stimulus: As an optimal algorithm drawn through the first year study, the vibratory stimulus is applied 10 times for 15 days (a 5-minute stimulus is applied two times a day for 10 days, and it is composed of repeated 15-second vibratory and 15-second non-vibratory stimulus with a strength of 3.3V).

ELIGIBILITY:
Inclusion Criteria

* A person who has at least 20 natural teeth, including the first molars (including fixed prostheses and implants, excluding removable prostheses)
* A person who has systemic health, including controlled hypertension/hypotension and diabetes patients
* An elderly person who has been diagnosed with normal cognition or mild cognitive impairment in a neuropsychological test and CERAD clinical evaluation (refer to separate inclusion criteria)

Exclusion Criteria

* A person who has medical history of nervous system disease
* A person who is has ever been allergic to resin
* A person who has untreated periodontal disease and/or severely loose teeth
* A person who has a medical treatment history of temporomandibular disorders, who has an occurrence of stomatitis once or more per month within the last 6 months, or who currently has stomatitis
* A person who is receiving or has received treatment for major mental diseases such as dementia, major depression, or mania based on the DSM-IV diagnosis
* A person who has a medical disease that can have a serious effect on cognitive function or is taking related medicine
* A person who has a transplant that is electrically or mechanically operated or a cerebrovascular clip or who has claustrophobia so that an MRI scan is impossible

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
cognitive function | 15 days
  Cambridge Neuropsychological Test Automated Battery (CANTAB, Cambridge Cognition, Cambridge, United Kingdom) (Sahgal, et al., 1992; Blackwell, et al., 2004; O'Connell, et al., 2004; Junkkila, Oja, Laine, & Karrasch, 2012)
  1. Paired Associates Learning (PAL) : Memory function
  2. Spatial Working Memory (SWM): frontal-executive function
  3. Stockings Of Cambridge (SOC): spatial planning ability and problem-solving ability

SECONDARY OUTCOMES:
quantitative electroencephalography (QEEG) and event-related potentials (ERPs) | 15 days
  : Based on a significant reduction of the relative power of α-wave (8-13Hz) and significant increase of the relative power of β-wave (13-30Hz)
  - Short-term and long-term ERP changes caused by oral vibratory stimulus: Change of amplitude and latency period of P300, the ERP component related to attention
functional magnetic resonance imaging (fMRI) | 15 days
  Assessing what difference the activated areas show compared to the results of the previous studies that identified the activated parts after masticatory activities when only oral vibratory stimulus is given without masticatory activities
masticatory ability | 15 days
  Unilateral maximal bite force is measured with a simple bite force gauge with a stick form (GM 10 occlusal force-meter: Nagano Keiki C., LTD, Japan). This is measured three times in a place where the subject feels at ease.
  * Maximum bite force: Numeric difference before and after the application of vibratory stimulus
  * Evaluation of masticatory ability: The change of Shape and color difference ofin gum before and after the application of vibratory stimulus
salivary secretion | 15 days
  * Evaluation of salivary secretion amount: mL per unit time (min) of saliva collected before and after the application of vibratory stimulus
  * Evaluation of compliance: The measurement of Tthe number of performances ofperforming the oral vibratory stimulus for 15 days for two times/day

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Jung Lee, Principal Investigator — Seoul National University Bundang Hospital

REFERENCES:
- [Background] Paganini-Hill A, White SC, Atchison KA. Dental health behaviors, dentition, and mortality in the elderly: the leisure world cohort study. J Aging Res. 2011;2011:156061. doi: 10.4061/2011/156061. Epub 2011 Jun 15. PMID 21748004
- [Background] Shimazaki Y, Soh I, Saito T, Yamashita Y, Koga T, Miyazaki H, Takehara T. Influence of dentition status on physical disability, mental impairment, and mortality in institutionalized elderly people. J Dent Res. 2001 Jan;80(1):340-5. doi: 10.1177/00220345010800010801. PMID 11269726